CLINICAL TRIAL: NCT05004337
Title: Verification of Risk Assignment for Whole Chromosome Using SNP-based NIPT in Vanishing Twin Pregnancies (VANISH)
Brief Title: Verification of Risk Assignment for Whole Chromosome Using SNP-based NIPT in Vanishing Twin Pregnancies
Acronym: VANISH
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-050-NPT
Record Dates: First submitted 2021-07-28; First posted 2021-08-13 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Vanishing Twin; Trisomy 21; Trisomy 13; Trisomy 18
MeSH Terms: conditions — Down Syndrome; Trisomy 13 Syndrome; Trisomy 18 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pregnancy blood samples from vanishing twin pregnancies and buccal samples from born babies in participating pregnancies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to collect blood samples from women carrying a vanishing twin pregnancy to further develop Natera's non-invasive prenatal screening test to provide information about possible chromosomal conditions for the living twin

ELIGIBILITY:
Inclusion Criteria:

* Women with either ultrasound-documented dizygotic (DZ) twin pregnancy or those whose Panorama Test™ results suggest increased risk for vanishing twin

Exclusion Criteria:

* Monozygotic twin pregnancy
* Non twin pregnancy
* Maternal history of bone marrow or organ transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women carrying a vanishing twin pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Develop a new algorithm and methodology that will measure fetal fraction and distinguish between the DT (demised/non-viable twin) and living twin (LT) in dizygotic twins (DZ) with a single LT. | 2 years
  A new algorithm will be written to analyze the serial research blood samples to return a fetal fraction of each twin, and identify which twin is the DT verses the LT. The fetal fraction measurement will be a percentage, and it will be measurable, or not measurable for each sample.
The accuracy of the new algorithm to determine which of the signals in the Panorama samples correspond to the LT versus the DT. | 2 Years
  Each complete participant in the study will have multiple maternal blood samples collected, and a child buccal swab. This outcome will use genetic analysis to reflect for each participant if the algorithm correctly or incorrectly identified the LT versus the DT. Accuracy, defined as the number of VT pairs correctly identified as the LT and DT, divided by the total number of VT pairs, will be calculated.

SECONDARY OUTCOMES:
The accuracy of the updated algorithm for the assignment of risk for trisomy 21/18/13 for the LT in DZ twins with a single LT. | 3 Years
  If a sufficient number of trisomy 21/18/13 cases are observed among any of the cases, assess the accuracy of the updated algorithm to correctly determine whether the LT or DT is aneuploidy. Point estimates and 95% confidence intervals for the specificity for the aneuploidy algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Vivienne Souter, MD, Study Chair — Natera, Inc.
Locations (21):
- United States (21):
  - Center for Fetal Medicine & Women's Ultrasound, Los Angeles, California
  - Stanford, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Yale, New Haven, Connecticut
  - Christiana Care, Newark, Delaware
  - Emerald Coast ObGyn, Panama City, Florida
  - University of Kansas, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Beaumont, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack, Neptune City, New Jersey
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - NYU Long Island, Mineola, New York
  - NYU Langone, New York, New York
  - Icahn School of Medicine at Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cedar Health Research, Irving, Texas